CLINICAL TRIAL: NCT07366749
Title: The Acute Effects of a Urate-lowering Probiotic Food Supplement/Bacterial Therapeutic on Small Intestinal Transcriptomics and Glycomics in Healthy Subjects
Brief Title: Acute Effects of a Urate-lowering Bacterial Therapeutic on Small Intestinal Transcriptomics and Glycomics in Healthy Subjects
Acronym: Bugs4U-MoA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: University of Copenhagen (Other); European Innovation Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2025-07972-01
Record Dates: First submitted 2026-01-09; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Hyperuricemia, Gout
Keywords: probiotics; gut microbiome; small intestine; transcriptomics; glycomics; urate metabolism
MeSH Terms: conditions — Hyperuricemia; Gout | interventions — beta-Glucans

STUDY DESIGN:
Intervention Model Description: Each participant receives all three interventions in a randomly assigned order. A minimum of 10 days separates each intervention period. This is intended to allow the gut to return to a baseline state and minimize carryover effects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotic (BEO001) (Active Comparator): Participants receive the BEO001 probiotic powder, which contains two probiotic strains
  Interventions: Dietary Supplement: BEO001 Probiotic
- Synbiotic (BEO001 + Beta-Glucan) (Active Comparator): Participants receive the BEO001 probiotic powder plus beta-glucan fiber powder.
  Interventions: Dietary Supplement: BEO001 Probiotic + Beta-Glucan
- Placebo (Placebo Comparator): Participants receive placebo powder.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: BEO001 Probiotic — A mixture of two probiotic strains. Total dose ≥5x10^10 CFU of each strain per intervention day. Administered as a powder mixed with water, consumed in several portions.
  Arms: Probiotic (BEO001)
Dietary Supplement: BEO001 Probiotic + Beta-Glucan — The BEO001 probiotic (as above) co-administered with 3g of a food-grade beta-glucan fiber. Both are powders mixed with water.
  Arms: Synbiotic (BEO001 + Beta-Glucan)
Dietary Supplement: Placebo — Powder without the active probiotic strains or beta-glucan
  Arms: Placebo

SUMMARY:
This is a pilot study investigating how a novel probiotic supplement (BEO001), with and without a dietary fiber (beta-glucan), affects the lining of the small intestine in healthy people. The main goal is to see if a single dose of the probiotic changes gene activity (transcriptomics) and sugar molecule patterns (glycomics) in the gut. Eight participants will take three different treatments (placebo, probiotic alone, probiotic with fiber) in a random order, with at least 10 days between each. A gastroscopy to collect small intestinal tissue samples (biopsies) is performed the morning after each treatment. Blood and breath samples are also collected at these visits to explore effects on metabolism and inflammation. To understand how different sampling methods compare, participants collect stool samples and simple rectal swabs at home before any treatment. Researchers analyze the sugar molecules and bacteria in these samples, then compare them to each other and to the gut tissue samples collected after treatment. This helps determine if easier-to-collect samples can provide similar information to gut biopsies. The study also aims to combine all data (including genetics and diet) to identify key targets for future research and to attempt to grow 'mini-gut' organoids from the biopsies. The results will help design larger future studies in people with high uric acid levels.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Age 18-60 years.
* BMI 18.5 - 29.9 kg/m².
* Willing to avoid probiotics, fermented foods, and maintain stable diet/lifestyle for the study duration.

Exclusion Criteria:

* Chronic GI, inflammatory, metabolic (including renal), or significant psychiatric disease.
* Acute infection/allergy within 2 weeks.
* Regular use of NSAIDs, antibiotics, steroids, immunomodulators.
* Alcohol >9 units/week.
* Use of recreational drugs, tobacco, or nicotine.
* Known allergy to local anesthetics or sedatives for gastroscopy.
* Bleeding disorder or use of anticoagulants.
* Use of probiotics or antibiotics within 4 weeks prior.
* Pregnancy, breastfeeding, or planning pregnancy.
* Any condition deemed by investigator to compromise safety or data integrity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in small intestinal transcriptomic profile after BEO001 intake | ~12-16 hours post-dose (at the gastroscopy visit).
  Gene expression profile (analyzed by RNA sequencing) in duodenal mucosal biopsies collected the morning after a single evening dose of BEO001 probiotic. Comparison is made between intervention visits (BEO001 vs. placebo).

SECONDARY OUTCOMES:
Change in small intestinal transcriptomic profile after BEO001+beta-glucan intake. | ~12-16 hours post-dose
  Gene expression profile in duodenal biopsies after a single evening dose of BEO001 with beta-glucan. Comparison is made between intervention visits (BEO001+beta-glucan vs. placebo).
Change in small intestinal glycomic profile after BEO001 intake | ~12-16 hours post-dose.
  N- and O-glycan profiles (analyzed by LC-MS) in duodenal biopsies after a single evening dose of BEO001. Comparison is made between intervention visits (BEO001 vs. placebo).
Change in small intestinal glycomic profile after BEO001+beta-glucan intake. | ~12-16 hours post-dose
  N- and O-glycan profiles in duodenal biopsies after a single evening dose of BEO001 with beta-glucan. Comparison is made between intervention visits (BEO001 +beta-glucan vs. placebo).

OTHER OUTCOMES:
Change in small intestinal mucosal microbiome composition and function. | ~12-16 hours post-dose.
  Microbial community profile and functional gene content (shotgun metagenomics) in duodenal biopsies. Comparison is made between intervention visits (BEO001 ± beta-glucan vs. placebo).
Change in blood urate concentrations | ~12-16 hours post-dose
  Levels of urate in blood . Comparison is made between intervention visits (BEO001 ± beta-glucan vs. placebo).
Change in blood creatinine | ~12-16 hours post-dose
  Levels of creatinine in blood . Comparison is made between intervention visits (BEO001 ± beta-glucan vs. placebo).
Change in blood metabolites and enzymes related to urate and inflammation. | ~12-16 hours post-dose.
  Concentrations of targeted metabolites and enzymes (including short-chain fatty acids) in blood. Comparison is made between intervention visits (BEO001 ± beta-glucan vs. placebo).
Change in Liver enzyme concentrations | ~12-16 hours post-dose.
  Levels of standard liver function enzymes (e.g., ALT, AST) in blood. Comparison is made between intervention visits (BEO001 ± beta-glucan vs. placebo).
Change in blood lipid profile. | ~12-16 hours post-dose
  Standard lipid panel measurements in blood. Comparison is made between intervention visits (BEO001 ± beta-glucan vs. placebo).
Change in the blood level of certain inflammatory cytokines | ~12-16 hours post-dose.
  Levels of certain inflammatory cytokines in blood will be measured. Comparison is made between intervention visits (BEO001 ± beta-glucan vs. placebo).
Change in blood level of C-reactive protein (hsCRP) | ~12-16 hours post-dose
  Levels of high-sensitivity C-reactive protein (hsCRP) in blood. Comparison is made between intervention visits (BEO001 ± beta-glucan vs. placebo).
Change in blood plasma glycomic profile | ~12-16 hours post-dose.
  N-glycan profile of total plasma proteins. Comparison is made between intervention visits (BEO001 ± beta-glucan vs. placebo).
Change in breath volatile organic compounds (VOCs). | ~12-16 hours post-dose.
  Profile of VOCs related to metabolism and inflammation in exhaled breath. Comparison is made between intervention visits (BEO001 ± beta-glucan vs. placebo).
Difference in glycomic profiles across biological sample types. | Rectal/faecal: Baseline (pre-intervention). Biopsies: ~12-16 hours post-dose.
  Comparison of glycomics profiles from baseline rectal swabs, baseline faecal samples, and post-intervention intestinal biopsies.
Difference in microbiome across biological sample types | Rectal/faecal: Baseline (pre-intervention). Biopsies: ~12-16 hours post-dose.
  Comparison of microbiome composition and function from baseline rectal swabs, baseline faecal samples, and post-intervention intestinal biopsies.
Correlation between outcomes and baseline characteristics. | Baseline characteristics (single measurement) correlated with outcomes measured ~12-16 hours post-dose.
  Analysis of associations between selected outcomes and screening/baseline characteristics (microbiome, metabolomics, glycomics, dietary patterns, genetic factors).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Brummer, MD, PhD, Study Director — Örebro universitet
Locations (1):
- Örebro University, Campus USO, School of medical sciences, Örebro, Örebro Lan, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
According to Swedish ethics regulations, IPD cannot be shared without an approved ethics application from the National Swedish Ethics Authority. An ethical permit can only be obtained for research being conducted within Sweden.